CLINICAL TRIAL: NCT06490159
Title: Predicting Peripheral Neuropathy of Paclitaxel in Second-line Chemotherapy for Gastric Cancer
Brief Title: Predicting Peripheral Neuropathy of Paclitaxel for Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/SLCGC-AE
Record Dates: First submitted 2024-06-16; First posted 2024-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Chemotherapy-induced Peripheral Neuropathy; Paclitaxel; Ramucirumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Ramucirumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample before second-line chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with peripheral neuropathy of paclitaxel in second-line chemotherapy for gastric cancer: A panel of microRNA, whose expression level is tested exosomal microRNA from blood sample before second-line chemotherapy with reverse transcriptase quantitative polymerase chain reaction (RT-qPCR)
  Interventions: Drug: Paclitaxel
- Patients without peripheral neuropathy of paclitaxel in second-line chemotherapy for gastric cancer: A panel of microRNA, whose expression level is tested exosomal microRNA from blood sample before second-line chemotherapy with reverse transcriptase quantitative polymerase chain reaction (RT-qPCR)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Gastric cancer second-line chemotherapy
  Other Names: Ramucirumab

SUMMARY:
Although advances in chemotherapy have improved the prognosis of gastric cancer patients, many patients still suffer from adverse events. Therefore, it is necessary to establish personalized treatment by identifying patients at high risk for side effects. Although paclitaxel-based therapy is the standard second-line treatment, peripheral neuropathy is a troublesome adverse event. The purpose of this study is to establish a liquid biopsy assay to predict paclitaxel-induced peripheral neuropathy in gastric cancer patients.

DETAILED DESCRIPTION:
Paclitaxel-based therapy is the standard second-line treatment for gastric cancer patients, but approximately 30-40% of patients develop peripheral neuropathy that interferes with daily life, and about 10% develop severe grade 3 peripheral neuropathy. Particularly severe side effects can cause patients to lose strength, forcing them to discontinue treatment, and thus losing the opportunity to receive other treatments that were originally expected to have a therapeutic effect. This study aims to predict peripheral neuropathy in the side effects of second-line treatment (paclitaxel plus ramucirumab) in patients with gastric cancer using liquid biopsies (small RNA). If patients at high risk for side effects can be predicted prior to treatment, high-risk patients can be offered drug reductions or other chemotherapy options. The aim of this study is to predict peripheral neuropathy of paclitaxel in second-line chemotherapy for gastric cancer by liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. unresectable or recurrent Gastric cancer (GC) histologically confirmed to be primary adenocarcinoma of the stomach.
2. age over 20 years.
3. Eastern Cooperative Oncology Group performance status score of 0-2.
4. written informed consent following full study information is provided to the patient.
5. progression or intolerance for first-line chemotherapy comprising fluorinated pyrimidine and platinum anticancer drugs (cisplatin or oxaliplatin) for advanced GC.
6. presence of evaluable lesions as confirmed using a computed tomography (CT) or magnetic resonance imaging.

Exclusion Criteria:

1. Patients with a life expectancy of shorter than 3 months
2. Patients with severe complications (angina pectoris, myocardial infarction, or arrhythmia) or uncontrollable diabetes mellitus, blood hypertension, or bleeding tendency.
3. Patients with a history of serious allergic reactions or serious drug allergy.
4. Patients with a clinically relevant mental disorder that prohibits response to questionnaires.
5. Patients for whom the attending physician considered that enrollment in the study is inappropriate.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients need second-line chemotherapy with unresectable or recurrent Gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of peripheral neuropathy | 1 year
  The standard approach to treatment-related adverse events that occur during anticancer treatment is the Common Terminology Criteria for Adverse Events (CTCAE), which is maintained by the US National Cancer Institute.

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Takiguchi, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- Kawasaki Medical University, Kurashiki, Okayama-ken, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Ajani JA, D'Amico TA, Bentrem DJ, Chao J, Cooke D, Corvera C, Das P, Enzinger PC, Enzler T, Fanta P, Farjah F, Gerdes H, Gibson MK, Hochwald S, Hofstetter WL, Ilson DH, Keswani RN, Kim S, Kleinberg LR, Klempner SJ, Lacy J, Ly QP, Matkowskyj KA, McNamara M, Mulcahy MF, Outlaw D, Park H, Perry KA, Pimiento J, Poultsides GA, Reznik S, Roses RE, Strong VE, Su S, Wang HL, Wiesner G, Willett CG, Yakoub D, Yoon H, McMillian N, Pluchino LA. Gastric Cancer, Version 2.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 Feb;20(2):167-192. doi: 10.6004/jnccn.2022.0008. PMID 35130500
- [Background] Park SR, Kim MJ, Nam BH, Kim CG, Lee JY, Cho SJ, Kong SY, Park YI. A randomised phase II study of continuous versus stop-and-go S-1 plus oxaliplatin following disease stabilisation in first-line chemotherapy in patients with metastatic gastric cancer. Eur J Cancer. 2017 Sep;83:32-42. doi: 10.1016/j.ejca.2017.06.008. Epub 2017 Jul 14. PMID 28711577
- [Background] Shitara K, Lordick F, Bang YJ, Enzinger P, Ilson D, Shah MA, Van Cutsem E, Xu RH, Aprile G, Xu J, Chao J, Pazo-Cid R, Kang YK, Yang J, Moran D, Bhattacharya P, Arozullah A, Park JW, Oh M, Ajani JA. Zolbetuximab plus mFOLFOX6 in patients with CLDN18.2-positive, HER2-negative, untreated, locally advanced unresectable or metastatic gastric or gastro-oesophageal junction adenocarcinoma (SPOTLIGHT): a multicentre, randomised, double-blind, phase 3 trial. Lancet. 2023 May 20;401(10389):1655-1668. doi: 10.1016/S0140-6736(23)00620-7. Epub 2023 Apr 15. PMID 37068504
- [Background] Zhang J, Gao HF, Yang C, Zhu T, Ji F, Yang M, Zhang L, Li J, Cheng M, Zhang T, Shen B, Chen Y, Wang K. Prevention of taxane-associated acute pain syndrome with etoricoxib for patients with breast cancer: A phase II randomised trial. Eur J Cancer. 2022 Aug;171:150-160. doi: 10.1016/j.ejca.2022.05.019. Epub 2022 Jun 17. PMID 35724467
- [Background] Hirata K, Hamamoto Y, Ando M, Imamura CK, Yoshimura K, Yamazaki K, Hironaka S, Muro K. Weekly paclitaxel plus ramucirumab versus weekly nab-paclitaxel plus ramucirumab for unresectable advanced or recurrent gastric cancer with peritoneal dissemination refractory to first-line therapy-the P-SELECT trial (WJOG10617G)-a randomised phase II trial by the West Japan Oncology Group. BMC Cancer. 2020 Jun 12;20(1):548. doi: 10.1186/s12885-020-07047-1. PMID 32532230
- [Background] Hershman DL, Weimer LH, Wang A, Kranwinkel G, Brafman L, Fuentes D, Awad D, Crew KD. Association between patient reported outcomes and quantitative sensory tests for measuring long-term neurotoxicity in breast cancer survivors treated with adjuvant paclitaxel chemotherapy. Breast Cancer Res Treat. 2011 Feb;125(3):767-74. doi: 10.1007/s10549-010-1278-0. Epub 2010 Dec 3. PMID 21128110
- [Background] Mo H, Yan X, Zhao F, Teng Y, Sun X, Lv Z, Cao M, Zhao J, Song G, Pan B, Li H, Zhai J, Xu B, Ma F. Association of Taxane Type With Patient-Reported Chemotherapy-Induced Peripheral Neuropathy Among Patients With Breast Cancer. JAMA Netw Open. 2022 Nov 1;5(11):e2239788. doi: 10.1001/jamanetworkopen.2022.39788. PMID 36322088
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Battaglini E, Goldstein D, Grimison P, McCullough S, Mendoza-Jones P, Park SB. Chemotherapy-Induced Peripheral Neurotoxicity in Cancer Survivors: Predictors of Long-Term Patient Outcomes. J Natl Compr Canc Netw. 2021 Jul 28;19(7):821-828. doi: 10.6004/jnccn.2021.7026. PMID 34340206
- [Background] Ma S, Zhou M, Xu Y, Gu X, Zou M, Abudushalamu G, Yao Y, Fan X, Wu G. Clinical application and detection techniques of liquid biopsy in gastric cancer. Mol Cancer. 2023 Jan 11;22(1):7. doi: 10.1186/s12943-023-01715-z. PMID 36627698
- [Background] Zhou X, Jia Y, Mao C, Liu S. Small extracellular vesicles: Non-negligible vesicles in tumor progression, diagnosis, and therapy. Cancer Lett. 2024 Jan 1;580:216481. doi: 10.1016/j.canlet.2023.216481. Epub 2023 Nov 15. PMID 37972701
- [Background] Tovar-Camargo OA, Toden S, Goel A. Exosomal microRNA Biomarkers: Emerging Frontiers in Colorectal and Other Human Cancers. Expert Rev Mol Diagn. 2016;16(5):553-67. doi: 10.1586/14737159.2016.1156535. Epub 2016 Mar 16. PMID 26892862
- [Background] Balusu S, Van Wonterghem E, De Rycke R, Raemdonck K, Stremersch S, Gevaert K, Brkic M, Demeestere D, Vanhooren V, Hendrix A, Libert C, Vandenbroucke RE. Identification of a novel mechanism of blood-brain communication during peripheral inflammation via choroid plexus-derived extracellular vesicles. EMBO Mol Med. 2016 Oct 4;8(10):1162-1183. doi: 10.15252/emmm.201606271. Print 2016 Oct. PMID 27596437
- [Background] Yu W, Hurley J, Roberts D, Chakrabortty SK, Enderle D, Noerholm M, Breakefield XO, Skog JK. Exosome-based liquid biopsies in cancer: opportunities and challenges. Ann Oncol. 2021 Apr;32(4):466-477. doi: 10.1016/j.annonc.2021.01.074. Epub 2021 Feb 4. PMID 33548389
- [Background] Shigeyasu K, Toden S, Zumwalt TJ, Okugawa Y, Goel A. Emerging Role of MicroRNAs as Liquid Biopsy Biomarkers in Gastrointestinal Cancers. Clin Cancer Res. 2017 May 15;23(10):2391-2399. doi: 10.1158/1078-0432.CCR-16-1676. Epub 2017 Jan 31. PMID 28143873
- [Background] Jung G, Hernandez-Illan E, Moreira L, Balaguer F, Goel A. Epigenetics of colorectal cancer: biomarker and therapeutic potential. Nat Rev Gastroenterol Hepatol. 2020 Feb;17(2):111-130. doi: 10.1038/s41575-019-0230-y. Epub 2020 Jan 3. PMID 31900466
- [Background] Tanioka H, Nagasaka T, Uno F, Inoue M, Okita H, Katata Y, Kanzaki H, Kuramochi H, Satake H, Shindo Y, Doi A, Nasu J, Yamashita H, Yamaguchi Y. The relationship between peripheral neuropathy and efficacy in second-line chemotherapy for unresectable advanced gastric cancer: a prospective observational multicenter study protocol (IVY). BMC Cancer. 2019 Oct 11;19(1):941. doi: 10.1186/s12885-019-6163-6. PMID 31604467
- [Background] Shitara K, Takashima A, Fujitani K, Koeda K, Hara H, Nakayama N, Hironaka S, Nishikawa K, Makari Y, Amagai K, Ueda S, Yoshida K, Shimodaira H, Nishina T, Tsuda M, Kurokawa Y, Tamura T, Sasaki Y, Morita S, Koizumi W. Nab-paclitaxel versus solvent-based paclitaxel in patients with previously treated advanced gastric cancer (ABSOLUTE): an open-label, randomised, non-inferiority, phase 3 trial. Lancet Gastroenterol Hepatol. 2017 Apr;2(4):277-287. doi: 10.1016/S2468-1253(16)30219-9. Epub 2017 Jan 19. PMID 28404157
- [Background] Bando H, Shimodaira H, Fujitani K, Takashima A, Yamaguchi K, Nakayama N, Takahashi T, Oki E, Azuma M, Nishina T, Hironaka S, Komatsu Y, Shitara K. A phase II study of nab-paclitaxel in combination with ramucirumab in patients with previously treated advanced gastric cancer. Eur J Cancer. 2018 Mar;91:86-91. doi: 10.1016/j.ejca.2017.11.032. Epub 2018 Jan 30. PMID 29353164
- [Background] Xu RH, Zhang Y, Pan H, Feng J, Zhang T, Liu T, Qin Y, Qin S, Yin X, Liu B, Ba Y, Yang N, Voon PJ, Tanasanvimon S, Zhou C, Zhang WL, Shen L. Efficacy and safety of weekly paclitaxel with or without ramucirumab as second-line therapy for the treatment of advanced gastric or gastroesophageal junction adenocarcinoma (RAINBOW-Asia): a randomised, multicentre, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2021 Dec;6(12):1015-1024. doi: 10.1016/S2468-1253(21)00313-7. Epub 2021 Oct 7. PMID 34626550
- [Background] Moehler M, Xiao H, Blum SI, Elimova E, Cella D, Shitara K, Ajani JA, Janjigian YY, Garrido M, Shen L, Yamaguchi K, Liu T, Schenker M, Kowalyszyn R, Bragagnoli AC, Bruges R, Montesarchio V, Pazo-Cid R, Hunter S, Davenport E, Wang J, Kondo K, Li M, Wyrwicz L. Health-Related Quality of Life With Nivolumab Plus Chemotherapy Versus Chemotherapy in Patients With Advanced Gastric/Gastroesophageal Junction Cancer or Esophageal Adenocarcinoma From CheckMate 649. J Clin Oncol. 2023 Dec 10;41(35):5388-5399. doi: 10.1200/JCO.23.00170. Epub 2023 Sep 15. PMID 37713657
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Kang YK, Chen LT, Ryu MH, Oh DY, Oh SC, Chung HC, Lee KW, Omori T, Shitara K, Sakuramoto S, Chung IJ, Yamaguchi K, Kato K, Sym SJ, Kadowaki S, Tsuji K, Chen JS, Bai LY, Oh SY, Choda Y, Yasui H, Takeuchi K, Hirashima Y, Hagihara S, Boku N. Nivolumab plus chemotherapy versus placebo plus chemotherapy in patients with HER2-negative, untreated, unresectable advanced or recurrent gastric or gastro-oesophageal junction cancer (ATTRACTION-4): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):234-247. doi: 10.1016/S1470-2045(21)00692-6. Epub 2022 Jan 11. PMID 35030335
- [Background] Hironaka S, Ueda S, Yasui H, Nishina T, Tsuda M, Tsumura T, Sugimoto N, Shimodaira H, Tokunaga S, Moriwaki T, Esaki T, Nagase M, Fujitani K, Yamaguchi K, Ura T, Hamamoto Y, Morita S, Okamoto I, Boku N, Hyodo I. Randomized, open-label, phase III study comparing irinotecan with paclitaxel in patients with advanced gastric cancer without severe peritoneal metastasis after failure of prior combination chemotherapy using fluoropyrimidine plus platinum: WJOG 4007 trial. J Clin Oncol. 2013 Dec 10;31(35):4438-44. doi: 10.1200/JCO.2012.48.5805. Epub 2013 Nov 4. PMID 24190112
- [Background] Shitara K, Doi T, Dvorkin M, Mansoor W, Arkenau HT, Prokharau A, Alsina M, Ghidini M, Faustino C, Gorbunova V, Zhavrid E, Nishikawa K, Hosokawa A, Yalcin S, Fujitani K, Beretta GD, Cutsem EV, Winkler RE, Makris L, Ilson DH, Tabernero J. Trifluridine/tipiracil versus placebo in patients with heavily pretreated metastatic gastric cancer (TAGS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1437-1448. doi: 10.1016/S1470-2045(18)30739-3. Epub 2018 Oct 21. PMID 30355453
- [Background] Shitara K, Bang YJ, Iwasa S, Sugimoto N, Ryu MH, Sakai D, Chung HC, Kawakami H, Yabusaki H, Lee J, Saito K, Kawaguchi Y, Kamio T, Kojima A, Sugihara M, Yamaguchi K; DESTINY-Gastric01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Gastric Cancer. N Engl J Med. 2020 Jun 18;382(25):2419-2430. doi: 10.1056/NEJMoa2004413. Epub 2020 May 29. PMID 32469182
- [Background] Cavaletti G, Zanna C. Current status and future prospects for the treatment of chemotherapy-induced peripheral neurotoxicity. Eur J Cancer. 2002 Sep;38(14):1832-7. doi: 10.1016/s0959-8049(02)00229-0. No abstract available. PMID 12204664
- [Background] Park SB, Kwok JB, Asher R, Lee CK, Beale P, Selle F, Friedlander M. Clinical and genetic predictors of paclitaxel neurotoxicity based on patient- versus clinician-reported incidence and severity of neurotoxicity in the ICON7 trial. Ann Oncol. 2017 Nov 1;28(11):2733-2740. doi: 10.1093/annonc/mdx491. PMID 29117336
- [Background] Meregalli C, Fumagalli G, Alberti P, Canta A, Chiorazzi A, Monza L, Pozzi E, Carozzi VA, Blennow K, Zetterberg H, Cavaletti G, Marmiroli P. Neurofilament light chain: a specific serum biomarker of axonal damage severity in rat models of Chemotherapy-Induced Peripheral Neurotoxicity. Arch Toxicol. 2020 Jul;94(7):2517-2522. doi: 10.1007/s00204-020-02755-w. Epub 2020 Apr 24. PMID 32333051
- [Background] Sakai A, Saitow F, Maruyama M, Miyake N, Miyake K, Shimada T, Okada T, Suzuki H. MicroRNA cluster miR-17-92 regulates multiple functionally related voltage-gated potassium channels in chronic neuropathic pain. Nat Commun. 2017 Jul 5;8:16079. doi: 10.1038/ncomms16079. PMID 28677679
- [Background] Yi S, Yuan Y, Chen Q, Wang X, Gong L, Liu J, Gu X, Li S. Regulation of Schwann cell proliferation and migration by miR-1 targeting brain-derived neurotrophic factor after peripheral nerve injury. Sci Rep. 2016 Jul 6;6:29121. doi: 10.1038/srep29121. PMID 27381812
- [Background] Zhi WI, Dreyfus N, Lessing A, Galantino M, Piulson L, Kot KL, Li S, Bao T. Patient Characteristics Associated With Chemotherapy-Induced Peripheral Neuropathy Severity in a Phase II Clinical Trial: A Retrospective Analysis. Oncologist. 2023 Jul 5;28(7):604-608. doi: 10.1093/oncolo/oyad062. PMID 36972359
- [Background] Greenlee H, Hershman DL, Shi Z, Kwan ML, Ergas IJ, Roh JM, Kushi LH. BMI, Lifestyle Factors and Taxane-Induced Neuropathy in Breast Cancer Patients: The Pathways Study. J Natl Cancer Inst. 2016 Oct 28;109(2):djw206. doi: 10.1093/jnci/djw206. Print 2017 Feb. PMID 27794123
- [Background] Lee S, Ma C, Shi Q, Kumar P, Couture F, Kuebler P, Krishnamurthi S, Lewis D, Tan B, Goldberg RM, Venook A, Blanke C, O'Reilly EM, Shields AF, Meyerhardt JA. Potential Mediators of Oxaliplatin-Induced Peripheral Neuropathy From Adjuvant Therapy in Stage III Colon Cancer: Findings From CALGB (Alliance)/SWOG 80702. J Clin Oncol. 2023 Feb 10;41(5):1079-1091. doi: 10.1200/JCO.22.01637. Epub 2022 Nov 11. PMID 36367997